CLINICAL TRIAL: NCT04361175
Title: Cost Effectiveness Analysis for Induction of Ovulation in the Polycystic Ovary Syndrome by Letrozole Versus Clomiphene Citrate: A Randomised Controlled Trial
Brief Title: Cost Effectiveness Analysis for Induction of Ovulation in the Polycystic Ovary Syndrome by Letrozole Versus Clomiphene Citrate
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nora Fayek Zaki, Residant doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Induction of ovulation
Record Dates: First submitted 2020-04-12; First posted 2020-04-24 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- letrozole group (Experimental): letrozole group, Patients will receive 5 mg of letrozole oral tablets daily from day 2 of the cycle for 5 days for three successive cycles
  Interventions: Drug: Letrozole
- Clomiphene Citrate group (Experimental): Clomiphene Citrate group, Patients will receive 100 mg : Clomiphene Citrate daily starting on cycle day 2 for 5 days for three successive cycles
  Interventions: Drug: Clomiphine Citrate

INTERVENTIONS:
Drug: Letrozole — Each group will be followed up for ovulation by day 12 ovulation monitoring by Transvaginal ultrasound for mature griffian follicle and measure endometrial thickness and volume then day 21 test serum progesterone level to confirm ovulation and if pregnancy occurred confirm by serum pregnancy test at day 35 of the cycle and follow pregnancy till confirmed by fetal pulsation by ultrasound.
  Arms: letrozole group
Drug: Clomiphine Citrate — Clomiphine Citrate
  Arms: Clomiphene Citrate group

SUMMARY:
To evaluate cost effectiveness of Letrozole versus clomiphene citrate (CC) in induction of ovulation in patients with polycystic ovary syndrome.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common cause of infertility that affects 4% - 8% of reproductive-age females (Priya,M.R,2019).

Diagnosis of PCOS is very important for proper management. In literature, Rotterdam criteria are widely used for diagnosis and focus on polycystic ovarian morphology on ultrasound,a history of ovulatory disorders (oligo-anovulation), and clinical/biochemical signs of hyperandrogenism requiring two of three features after exclusion of other endocrinopathies (Wang,R,2017).

Although the syndrome is a complex reproductive-metabolic disorder, the hypothalamic-pituitary axis has been the target of first-line ovulation-induction therapy. Clomiphene citrate, a selective estrogen-receptor modulator that antagonizes the negative feedback of estrogen at the hypothalamus with a consequent increase in ovarian stimulation by endogenous gonadotropin, has been used for this indication for decades (Legro RS,2007).

Clomiphene citrate (CC) is still holding its place for ovulation induction being simple, safe, cheap and effective (Garg, N,2019).

However, clomiphene-resistance, i.e., failure to ovulate after receiving 150 mg/day for at least three cycles for five days per cycle affects 15% - 40% of patients with PCOS (Salaheldin,A.M,2016).

Aromatase inhibitors, which block estrogen synthesis, directly affect hypothalamic- pituitary-ovarian function and theoretically might increase pregnancy rates (Casper RF,2006).

Many tissues including the ovary (in premenopausal women), fat, muscle, breast and liver contain aromatase enzyme which controls the ﬁnal step in estrogen synthesis, It is responsible for aromatization of androstenedione and testosterone into estrone and estradiol, respectively. This process can be inhibited by administration of a third-generation aromatase inhibitor such as letrozole by >99% (Haynesa,B.P,2003).

Letrozole has become the first line drug for induction of ovulation in PCOS patients (Teede, H.J,2018).

ELIGIBILITY:
Inclusion criteria:

* Women with infertility secondary to PCOS according to ESHRE/ASRM (Rotterdam criteria) 2004. Patients have at least two of the following; clinical and/or biochemical hyperandrogenism, oligo-ovulation or anovulation, polycystic ovaries by sonography (Diagnosis of oligo-/anovulation will be based on a menstrual pattern of oligo-/amenorrhoea (cycle >35 days) and/or a low mid-luteal serum progesterone concentration. Hyperandrogenaemia will be diagnosed either clinically (acne/hirsutism) or biochemically (testosterone ≥2.5 nmol/l or free androgen index [FAI] ≥5). Ultrasound criteria will include ≥12 follicles (2-9 mm) and/or an ovarian volume of >10 ml).
* Age between 18 to 35 years with Body Mass Index (BMI) not more than 35 kg/m2, free of any medical disease and not receiving medications in the last 3 months.

Exclusion criteria:

* Patients with other causes of infertility, gross ovarian pathology diagnosed by ultrasound, previous tubal or ovarian surgery or laparoscopic ovarian drilling will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 212 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Ovulation detection by Trans-vaginal ultrasound in day 12 of menstrual cycle | Three months
  ovulation monitoring by Trans-vaginal ultrasound (Medison SonoACEX6 Soul Korea 2012 ) for mature GF in each group.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Casper RF, Mitwally MF. Review: aromatase inhibitors for ovulation induction. J Clin Endocrinol Metab. 2006 Mar;91(3):760-71. doi: 10.1210/jc.2005-1923. Epub 2005 Dec 29. PMID 16384846